CLINICAL TRIAL: NCT00576628
Title: A Single Arm Open Label Multicentre Study to Assess the Efficacy, Safety and Tolerability of Monthly Administration of Subcutaneous C.E.R.A. for the Treatment of Chronic Renal Anaemia in Pre-dialysis Patients, Not Currently Treated With ESA
Brief Title: A Study of Subcutaneous C.E.R.A. for the Treatment of Anemia in Pre-Dialysis Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20978
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- C.E.R.A (Experimental): Participants received methoxy polyethylene glycol-epoetin beta (Continuous Erythropoietin Receptor Activator [C.E.R.A]) subcutaneously every four weeks for 44 weeks. The participants received initial dose of 1.2 microgram per kilogram (mcg/kg) of C.E.R.A. Once the Hemoglobin (Hb) concentration was attained within the target range of 11.0 and 13.0 gram per deciliter (g/dL), the dose was adjusted to maintain the Hb concentration within the target range.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [C.E.R.A.]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [C.E.R.A.] — Recommended starting dose 1.2 micrograms/kg sc monthly

SUMMARY:
This single arm study will assess the efficacy, safety and tolerability of subcutaneous C.E.R.A. for correction of anemia and maintenance of hemoglobin levels in patients with chronic kidney disease who are not on dialysis and are not treated with ESA. Eligible patients will receive C.E.R.A. by monthly subcutaneous injections, dependent on body weight (with a recommended starting dose of 1.2 micrograms/kg). The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia, with no need for dialysis expected in next 3 months;
* adequate iron status.

Exclusion Criteria:

* previous epoetin therapy within 12 weeks prior to treatment;
* transfusion of red blood cells during 2 months prior to screening;
* significant acute or chronic bleeding such as overt gastrointestinal bleeding;
* hemolysis;
* folic acid and vitamin B 12 deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Russia (12):
  - Irkutsk
  - Khanty-Mansiysk
  - Moscow
  - Nizhny Novgorod
  - Omsk
  - Orenburg
  - Rostov-on-Don
  - Saint Petersburg
  - Saratov
  - Tyumen
  - Ufa
  - Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 133 eligible participants were enrolled in the study conducted from 8 May 2008 to 31 March 2010 across 19 centers in Russia.
Pre-assignment Details: Out of total 133 enrolled participants who met the eligibility criteria, eight participants did not receive active study drug and were not included in any analysis population.
Period: Overall Study
Arm/Group | C.E.R.A
Started | 125
Completed | 82
Not Completed | 43
Not completed — Adverse Event | 11
Not completed — Death | 2
Not completed — Failure to return | 1
Not completed — Refused Treatment | 8
Not completed — Pregnancy | 1
Not completed — RBC transfusion | 1
Not completed — Progression of Kidney Disease | 1
Not completed — Progression of Renal Failure | 1
Not completed — The patient move into other town | 1
Not completed — Transplantation | 1
Not completed — Dialysis | 15

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who received at least one dose of C.E.R.A. (Week 0) and for whom data for at least one follow-up variable were available.
Groups:
- C.E.R.A: Participants received C.E.R.A subcutaneously every four weeks for 44 weeks. The participants received initial dose of 1.2 mcg/kg of C.E.R.A. Once the Hb concentration was attained within the target range of 11.0 and 13.0 g/dL, the dose was adjusted to maintain the Hb concentration within the target range.
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (15.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hb Concentration g/dL Between Baseline and the Efficacy Evaluation Period
Description: The mean change in Hb concentration between Baseline and Efficacy Evaluation Period (EEP) was calculated by subtracting the baseline Hb concentration from the EEP Hb concentration. Each participant included in this analysis had at least 3 recorded Hb values during EEP, and these Hb values were combined using a time-adjusted average. The EEP was from Week 29 to Week 36.
Time Frame: Baseline (Week 0) and from Week 29 to Week 36
Population: The primary analysis was performed on per protocol (PP) population. The PP population included all treated participants (ITT participants) except those who had less than 3 recorded Hb values during EEP or with inadequate iron status during the EEP or missed administrations of C.E.R.A. during Week 28 to Week 36.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A
Number analyzed (Participants) | 66
g/dL | 1.75 (1.09)

2. Secondary Outcome: Percentage of Participants Maintaining Average Hb Concentration Within the Target Range of 11.0-13.0 g/dL Throughout the EEP
Description: Percentage of participants maintaining individual Hb concentration within the range of 11.0-13.0 g/dL was reported during EEP. The EEP was from Week 29 to Week 36.
Time Frame: From Week 29 to Week 36
Population: The primary analysis was performed on PP population. The PP population included all treated participants (ITT participants) except those who had less than 3 recorded Hb values during EEP or with inadequate iron status during the EEP or missed administrations of C.E.R.A. during Week 28 to Week 36.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 66
percentage of participants | 66.7 [54.0 to 77.8]

3. Secondary Outcome: Mean Time Spent in Target Hb Range of 11.0 -13.0 g/dL During the Efficacy Evaluation Period
Description: The number of days spent by participants with Hb in range of 11.30 -13.0 g/dL was calculated during the EEP and presented. The EEP comprised was from Week 29 to Week 36.
Time Frame: From Week 29 to Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C.E.R.A
Number analyzed (Participants) | 66
days | 37.4 (18.98)

4. Secondary Outcome: The Number of Participants Who Required Dose Adjustments During the Dose Titration Period
Description: The number of participants who required dose adjustments of C.E.R.A was reported during the Dose Titration Period (DTP). The DTP was from Week 0 to Week 28.
Time Frame: From Week 0 to Week 28 (DTP)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 66
participants | 61

5. Secondary Outcome: Time to Achievement of Response During the Efficacy Evaluation Period
Description: The time to achievement of response was defined as the time when the participants achieved Hb concentration within the target range of 11.0 to 13.0 g/dL during the EEP. The EEP was from Week 29 to Week 36.
Time Frame: From Week 29 to Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C.E.R.A
Number analyzed (Participants) | 66
days | 30.8 (27.21)

6. Secondary Outcome: Number of Participants With Red Blood Cells Transfusions.
Description: The number of participants who received at least 1 red blood cell (RBC) transfusion (packed RBC or whole blood) during the study was reported.
Time Frame: Up to Week 52
Population: The analysis was performed on safety population. The safety population included all the participants who received at least one dose of the trial medication and underwent a safety follow-up, whether withdrawn prematurely or not.
Measure: Number; unit: participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
participants | 1

7. Secondary Outcome: Mean Values of Laboratory Parameter : Hb Concentration
Description: The mean Hb concentration for each individual participant throughout the study was estimated. Summary data of mean values of Hb concentration at Week 0 (Baseline), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48 are presented.
Time Frame: Baseline (Week 0), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: The analysis was performed on safety population. The safety population included all the participants who received at least one dose of the trial medication and underwent a safety follow-up, whether withdrawn prematurely or not. The "n" represents the number of participants analyzed at a specified time point.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
g/dL
  Baseline, n = 125 | 10.0 (0.58)
  Week 8, n = 115 | 11.7 (1.26)
  Week 16, n = 104 | 12.2 (1.17)
  Week 24, n = 101 | 11.6 (1.12)
  Week 32, n = 90 | 12.0 (1.12)
  Week 40, n = 85 | 11.8 (1.14)
  Week 48, n = 82 | 11.6 (1.06)

8. Secondary Outcome: Mean Values of Laboratory Parameter : Hematocrit
Description: Hematocrit is a blood test that measures the percentage of the volume of whole blood that is made up of red blood cells (RBC). This measurement depends on the number of red blood cells and the size of red blood cells. The mean values of hematocrit for each individual participant were estimated throughout the study. Summary data of mean values of hematocrit at Week 0 (Baseline), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48 are presented.
Time Frame: Baseline (Week 0), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: fraction
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
fraction
  Baseline, n = 124 | 0.30 (0.03)
  Week 8, n = 112 | 0.34 (0.04)
  Week 16, n = 103 | 0.36 (0.04)
  Week 24, n = 101 | 0.34 (0.04)
  Week 32, n = 90 | 0.35 (0.04)
  Week 40; n = 85 | 0.35 (0.05)
  Week 48, n = 82 | 0.34 (0.04)

9. Secondary Outcome: Mean Values of Laboratory Parameters: Potassium and Phosphate Concentration
Description: The mean values of potassium and phosphate levels in serum for each individual participant were estimated throughout the study. Summary data of mean values of potassium and phosphate level in serum at Week 0 (Baseline), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48 are presented.
Time Frame: Baseline (Week 0), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimoles per litre
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
millimoles per litre
  Phosphate, Baseline, n = 124 | 1.5 (0.36)
  Phosphate, Week 8, n = 113 | 1.6 (0.38)
  Phosphate, Week 16, n = 102 | 1.5 (0.47)
  Phosphate, Week 24, n = 94 | 1.6 (0.37)
  Phosphate, Week 32, n = 85 | 1.6 (0.45)
  Phosphate, Week 40, n = 80 | 1.6 (0.46)
  Phosphate, Week 48, n = 79 | 1.6 (0.49)
  Potassium, Baseline, n = 125 | 5.1 (0.60)
  Potassium, Week 8, n=113 | 5.1 (0.66)
  Potassium, Week 16, n = 102 | 5.1 (0.59)
  Potassium, Week 24, n= 96 | 5.0 (0.75)
  Potassium, Week 32, n = 85 | 5.1 (0.59)
  Potassium, Week 40, n = 79 | 5.1 (0.56)
  Potassium, Week 48, n = 80 | 5.2 (0.76)

10. Secondary Outcome: Mean Values of Laboratory Parameter : Iron and Total Iron Binding Capacity
Description: The mean values of iron and total iron binding capacity (TIBC) for each individual participant were estimated throughout the study. Summary data of mean values of iron and TIBC at Week 0 (Baseline), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48 are presented.
Time Frame: Baseline (Week 0), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
micromoles/liter
  Iron, Baseline, n = 125 | 16.0 (5.35)
  Iron, Week 8, n = 113 | 14.0 (6.35)
  Iron, Week 16, n = 103 | 14.9 (6.25)
  Iron, Week 24, n = 96 | 15.9 (6.10)
  Iron, Week 32, n = 84 | 16.6 (6.22)
  Iron, Week 40, n = 79 | 15.7 (6.20)
  Iron, Week 48, n = 81 | 16.4 (5.83)
  TIBC, Baseline, n = 58 | 49.2 (15.46)
  TIBC, Week 8, n = 55 | 53.7 (13.57)
  TIBC, Week 16, n = 45 | 53.5 (13.67)
  TIBC, Week 24, n = 44 | 54.8 (13.71)
  TIBC, Week 32, n = 38 | 50.6 (11.93)
  TIBC, Week 40, n = 35 | 54.0 (13.35)
  TIBC, Week 48, n = 36 | 51.5 (12.17)

11. Secondary Outcome: Mean Values of Laboratory Parameter : Serum Creatinine
Description: The mean values of serum creatinine for each individual participant throughout the study were estimated. Summary data of mean values of serum creatinine at Week 0 (Baseline) and Week 32 are presented.
Time Frame: Baseline (Week 0), and Week 32
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micromoles/liter
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
micromoles/liter
  Creatinine, Baseline, n = 125 | 317.8 (145.41)
  Creatinine, Week 32, n = 84 | 361.3 (160.27)

12. Secondary Outcome: Mean Values of Laboratory Parameter: C Reactive Protein
Description: The mean values of C reactive protein (CRP) for each individual participant throughout the study were estimated. Summary data of mean values of CRP at Week 0 (Baseline), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48 are presented.
Time Frame: Baseline (Week 0), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per liter
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
milligrams per liter
  CRP, Baseline, n = 123 | 4.1 (10.36)
  CRP, Week 8, n = 109 | 6.0 (15.02)
  CRP, Week 16, n = 101 | 6.5 (15.14)
  CRP, Week 24, n = 94 | 6.2 (15.14)
  CRP, Week 32, n = 81 | 4.5 (7.72)
  CRP, Week 40, n = 76 | 3.8 (6.00)
  CRP, Week 48, n = 79 | 4.1 (6.69)

13. Secondary Outcome: Mean Values of Laboratory Parameter: Albumin and Transferrin Concentration
Description: The mean values of albumin and transferrin concentration for each individual participant throughout the study were estimated. Summary data of mean values of albumin and transferrin concentration at Week 0 (Baseline), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48 are presented.
Time Frame: Baseline (Week 0), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
grams per liter
  Albumin, Baseline, n = 125 | 41.0 (6.66)
  Albumin, Week 8, n = 111 | 40.5 (6.18)
  Albumin, Week 16, n = 98 | 41.5 (6.15)
  Albumin, Week 24, n = 96 | 40.9 (6.28)
  Albumin, Week 32, n = 84 | 42.4 (5.82)
  Albumin, Week 40, n = 80 | 41.3 (7.31)
  Albumin, Week 48, n = 81 | 40.7 (5.46)
  Transferrin, Baseline, n = 86 | 2.0 (0.60)
  Transferrin, Week 8, n = 74 | 2.1 (0.47)
  Transferrin, Week 16, n = 81 | 2.1 (0.41)
  Transferrin, Week 24, n = 73 | 2.2 (0.41)
  Transferrin, Week 32, n = 67 | 2.1 (0.40)
  Transferrin, Week 40, n = 59 | 2.1 (0.46)
  Transferrin, Week 48, n = 61 | 2.1 (0.36)

14. Secondary Outcome: Mean Values of Laboratory Parameter: Ferritin Concentration
Description: The mean values of ferritin concentration for each individual participant throughout the study were estimated. Summary data of mean values of ferritin concentration at Week 0 (Baseline), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48 are presented.
Time Frame: Baseline (Week 0), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
micrograms per liter
  Ferritin, Baseline, n = 125 | 231.6 (167.47)
  Ferritin, Week 8, n = 112 | 152.4 (135.20)
  Ferritin, Week 16, n = 102 | 149.3 (113.26)
  Ferritin, Week 24, n = 94 | 154.1 (116.87)
  Ferritin, Week 32, n = 79 | 171.8 (150.75)
  Ferritin, Week 40, n = 74 | 179.6 (167.06)
  Ferritin, Week 48, n = 75 | 187.0 (204.67)

15. Secondary Outcome: Mean Values of Laboratory Parameters: White Blood Cell and Thrombocyte Count
Description: The mean values of white blood cell (WBC) and thrombocyte count for each individual participant were estimated throughout the study. Summary data of mean values of WBC and thrombocyte count at Week 0 (Baseline), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48 are presented.
Time Frame: Baseline (Week 0), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
10^9 cells/liter
  WBC, Baseline, n = 125 | 7.1 (2.22)
  WBC, Week 8, n = 114 | 7.2 (2.13)
  WBC, Week 16, n = 103 | 7.1 (2.20)
  WBC, Week 24, n = 97 | 7.1 (1.79)
  WBC, Week 32, n = 86 | 7.2 (1.76)
  WBC, Week 40, n = 80 | 6.9 (1.45)
  WBC, Week 48, n = 81 | 6.6 (1.56)
  Thrombocyte, Baseline, n = 125 | 255.4 (75.12)
  Thrombocyte, Week 8, n = 110 | 240.2 (69.63)
  Thrombocyte, Week 16, n = 102 | 237.3 (70.46)
  Thrombocyte, Week 24, n = 97 | 237.2 (66.31)
  Thrombocyte, Week 32, n = 85 | 237.0 (72.07)
  Thrombocyte, Week 40, n = 80 | 226.1 (53.30)
  Thrombocyte, Week 48, n = 81 | 222.5 (58.92)

16. Secondary Outcome: Mean Values of Laboratory Parameters: Transferrin Saturation
Description: The mean values for transferrin saturation (TSAT) for each individual participant were estimated throughout the study. Summary data of mean values of TSAT at Week 0 (Baseline), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48 are presented.
Time Frame: Baseline (Week 0), Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | C.E.R.A
Number analyzed (Participants) | 125
percentage of saturation
  TSAT, Baseline, n = 125 | 32.1 (18.59)
  TSAT, Week 8, n = 113 | 25.7 (13.57)
  TSAT, Week 16, n = 103 | 27.8 (12.14)
  TSAT, Week 24, n = 96 | 30.1 (12.02)
  TSAT, Week 32, n = 84 | 32.1 (13.82)
  TSAT, Week 40, n = 79 | 30.0 (14.37)
  TSAT, Week 48, n = 81 | 32.7 (16.72)

17. Secondary Outcome: The Number of Participants Who Required Dose Adjustments During the Efficacy Evaluation Period
Description: The number of participants who required dose adjustments of C.E.R.A was reported during the EEP. EEP was from Week 29 to Week 36.
Time Frame: From Week 29 to Week 36 (EEP)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 66
participants | 34

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: An adverse event (AE) was defined as any unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily, whether or not considered related to the treatment. Adverse event was summarized in participants who have been treated with at least one dose of the trial medication.
Arm/Group | C.E.R.A
Serious Adverse Events (participants affected / at risk) | 31/125
Other Adverse Events (participants affected / at risk) | 52/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A (N=125)
Acute myocardial infarction (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Coma (Nervous system disorders) | 2
Diabetic autonomic neuropathy (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Thrombotic stroke (Nervous system disorders) | 1
Vascular encephalopathy (Nervous system disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 9
Renal impairment (Renal and urinary disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Haemodialysis (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A (N=125)
Hypertension (Vascular disorders) | 28
Influenza (Infections and infestations) | 13
Asthenia (General disorders) | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 8
Blood Pressure Increased (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.